CLINICAL TRIAL: NCT02288598
Title: Enhancing Speech Fluency With Non-invasive Brain Stimulation in Developmental Stuttering
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSD-IDREC-C2-2014-013
Record Dates: First submitted 2014-09-30; First posted 2014-11-11 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Stuttering; Fluency Disorders; Speech Disorders
Keywords: Stammering; Brain stimulation
MeSH Terms: conditions — Stuttering; Speech Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anodal TDCS (Experimental): Participants will receive anodal TDCS over the left inferior frontal cortex. TDCS will be delivered at 1milliampere (mA) intensity for 20 minutes during speech fluency training (5 consecutive days).
  Interventions: Device: Anodal TDCS; Behavioral: Fluency Training
- Sham TDCS (Sham Comparator): Participants will receive sham TDCS over the left inferior frontal cortex. Sham stimulation will involve 30 seconds stimulation at the beginning of the 20 minutes of speech fluency training (5 consecutive days).
  Interventions: Behavioral: Fluency Training

INTERVENTIONS:
Device: Anodal TDCS — 20 minutes 1mA anodal stimulation to left inferior frontal cortex. Cathode positioned on right supra-orbital ridge.
  Arms: Anodal TDCS
Behavioral: Fluency Training — Speech tasks will be completed using fluency-enhancing techniques: metronome-timed speech and auditory choral speech.

SUMMARY:
This study aims to test whether the addition of transcranial direct current stimulation (TDCS) to speech fluency training results in improvements in speech fluency in adults with developmental stuttering. Half of the participants will receive anodal TDCS on five consecutive days, the other half will receive a sham stimulation for the same amount of time.

DETAILED DESCRIPTION:
Studies using TDCS have shown improvements in motor performance, and in expressive language skills in clinical and healthy populations. The benefits of single sessions of TDCS are short-lived. However, stimulation over multiple sessions can increase and prolong learning effects that can persist for several weeks after the end of the stimulation period. We aim to target left hemisphere frontal regions involved in speech production with TDCS, and to pair this stimulation with speech fluency training.

ELIGIBILITY:
Inclusion Criteria:

* Native speaker of English.
* Right handed.
* Participant has moderate to severe Developmental Stuttering (Stammering)

Exclusion Criteria:

* Speech, language or communication disorder other than Developmental Stuttering.
* Sensory impairment (hearing loss or visual impairment)
* History of drug abuse.
* History of seizures
* History of a neurological or psychiatric illness.
* History of neurosurgical procedure.
* Currently taking certain prescription medications such as anti-depressants and anti-malarial medication (as these may lower the seizure threshold)

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-10; Primary Completion 2016-03-14 (Actual); Study Completion 2016-03-14 (Actual)

PRIMARY OUTCOMES:
Change from baseline proportion of stuttering in speech sample | 1 week post-treatment
  Quantitative measurement of stuttering
Change from baseline proportion of stuttering in speech sample | 6 weeks post-treatment
  Quantitative measurement of stuttering

SECONDARY OUTCOMES:
Change from baseline on the Stuttering Severity Instrument version 4 (SSI-4) | 1 week post-treatment
  Standardised assessment of frequency and duration of stuttering and associated physical concomitants
Change from baseline on the Stuttering Severity Instrument version 4 (SSI-4) | 6 weeks post-treatment
  Standardised assessment of frequency and duration of stuttering and associated physical concomitants
Change from baseline on Overall Assessment of Speaker's Experience of Stuttering (OASES) | 6 weeks post-treatment
  Standardised assessment of the functional impact of stuttering on a person's life

CONTACTS AND LOCATIONS:
Overall Officials: Kate Watkins, PhD, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, Oxford, United Kingdom

REFERENCES:
- See also: Speech and Brain Research Group, University of Oxford — http://www.psy.ox.ac.uk/research/speech-brain-research-group